CLINICAL TRIAL: NCT01028586
Title: A Phase III, Double-blind, Placebo-controlled Extension Trial to Investigate the Long-term Efficacy and Safety of Low (50 mg/Day) and High (100 mg/Day) Dose Safinamide, as add-on Therapy in Subjects With Early Idiopathic Parkinson's Disease Treated With a Stable Dose of a Single Dopamine Agonist
Brief Title: MOTION, Safinamide in Early Idiopathic Parkinson's Disease (IPD), as add-on to Dopamine Agonist (Extension of Trial 27918)
Acronym: MOTION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial is terminated due to a company decision to return all rights for Safinamide back to Newron Pharmaceuticals
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27938; IND: 63,901
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2012-08

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: Safinamide, MAO-B inhibitor
- Arm 2 (Active Comparator): Number of Cycles: until progression or unacceptable toxicity develops.
  Interventions: Drug: Safinamide, MAO-B inhibitor
- Arm 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Safinamide, MAO-B inhibitor — Safinamide, MAO-B inhibitor 50 mg: once-daily orally for 78 weeks in addition to their dose of DA-agonist.
  Arms: Arm 1
Drug: Safinamide, MAO-B inhibitor — Safinamide, MAO-B inhibitor 100 mg: once-daily orally for 78 weeks in addition to their dose of DA-agonist.
  Arms: Arm 2
Drug: Placebo — matching placebo tablets
  Arms: Arm 3

SUMMARY:
Parkinson's disease is a major neurodegenerative disorder in which there is a progressive loss of nigrostriatal dopaminergic neurons. The understanding that PD is a syndrome of dopamine (DA) deficiency led to the introduction in the clinical practice of L-dopa, a precursor of DA that crosses the blood brain barrier, and also to the use of selective inhibitors of MAO B, the major DA metabolising enzyme in man.

This is a double-blind, placebo-controlled, extension trial, parallel-group, randomised, multi-centre, multi national, Phase III trial, comparing two doses of safinamide (50 and 100 mg p.o. q.a.m.) versus placebo as add-on therapy to a stable dose of a single dopamine agonist in subjects with early idiopathic Parkinson's Disease.

The principal objective is to evaluate the time to first intervention, as some previous data suggested that safinamide may delay the need for further dopaminergic supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. The subject completed 24 weeks of Trial 27918.
2. The subject successfully completed all trial requirements in Trial 27918.
3. If female, they must be either post menopausal for at least 2 years, surgically sterilized or have undergone hysterectomy or, if of child bearing potential they must be willing to avoid pregnancy by using an adequate method of contraception as defined in the protocol for four weeks prior to, during and four weeks after the last dose of trial medication. For the purposes of this trial, women of childbearing potential are defined as: "All female subjects after puberty unless they are post-menopausal for at least two years, are surgically sterile or are sexually inactive".
4. Subject is willing and able to participate in the trial and has provided written, informed consent

Exclusion Criteria:

1. If female, the subject is pregnant or lactating.
2. The subject experienced a clinically significant adverse effect during trial 27918 that could put the subject at risk according to the investigator's opinion.
3. The subject has shown clinically significant deterioration during participation in Trial 27918.
4. Motor deterioration during trial 27918 that required upward titration of existing anti-parkinsonian medication or the initiation of an additional anti-parkinsonian medication.
5. The investigator deems it is not in the subject's best interest to participate to trial 27938
6. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Time from baseline to first intervention, i.e., change in the dose of Dopamine (DA) agonist, addition of another DA-agonist, levodopa, or other Parkinson Disease (PD) therapy, or discontinuation due to lack of efficacy | Week 78

SECONDARY OUTCOMES:
Proportion of subjects requiring intervention | Week 78
Unified Parkinson's Disease Rating Scale (UPDRS) Section III (motor) score change from baseline to week 78 | Week 78
Unified Parkinson's Disease Rating Scale (UPDRS) Section II (ADL) score change from baseline to week 78 | Week 78
Clinical Global impression (CGI) - Change scale score, change from Day 0 of Trial 27918 to week 78 | Week 78
Clinical Global impression (CGI) - Severity scale score change from baseline to week 78 | Week 78
EuroQoL 5D (EQ-5D) score change from baseline to week 78 | Week 78
Parkinson's Disease Questionnaire (PDQ-39) score change from baseline to week 78 | Week 78
Cogtest® PD battery test score change from baseline to week 78 | Week 78

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Willmer, MD, Study Director — EMD Serono
Locations (1):
- Enquire Central Contact, Geneva, Switzerland